CLINICAL TRIAL: NCT04799470
Title: Novel DBS Stimulation Patterns for Treatment of Parkinson's Disease - UNMC/Medtronic Collaborative Acute Feasibility Pilot
Brief Title: Novel DBS Stimulation Patterns for Treatment of Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0865-20-FB
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PD with DBS (Experimental): Patients with Parkinson's Disease who were implanted with Medtronic Percept PC for DBS and consent to participate in the study.
  Interventions: Device: Novel DBS stimulation patterns

INTERVENTIONS:
Device: Novel DBS stimulation patterns — Stimulation patterns

SUMMARY:
This is an open-label, non-randomized, proof-of-concept comparison of clinical vs. research stimulation patterns in patients with Parkinson's disease (PD) being treated with Deep Brain Stimulation (DBS) through the Medtronic Percept PC DBS device. The investigators hypothesize that stimulation patterns designed to better target excessive synchrony in a patient-tailored manner may result in more efficient and effective therapy with fewer side effects. Medtronic 3rd-generation sensing implantable neural stimulator, Percept PC, is FDA-approved for treating PD. The Percept PC device features BrainSense, the first and only available sensing technology for deep brain stimulation. BrainSense technology allows the device to capture and record brain signals (local field potentials, or LFP) using the brain-implanted DBS lead, while simultaneously delivering therapeutic stimulation. Investigators plan to enroll and complete investigations in 15 study subjects total, who have been previously implanted with the Medtronic Percept PC for the treatment of PD, and who are optimized for clinical stimulation and anti-Parkinsons medication. Investigations will be performed in UNMC Movement Disorders Clinic, UNMC Neurosurgery Lab, and UNO Biomechanics Research Building, Gait Lab. Subjects will receive research stimulation patterns and the effect on PD motor symptoms will be assessed via Unified Parkinsons Disease Rating Scale (UPDRS)-part III and gait measures. Videotaping of patient UPDRS-III testing and gait will be obtained.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by both motor and non-motor symptoms. Motor symptoms of PD include the clinical triad of tremor, rigidity, and bradykinesia, and typically lead to the initial diagnosis. While there is yet no cure for PD, medical and surgical therapies have been developed that effectively target the motor symptoms of PD. Patients with PD who demonstrate significant motor fluctuations and dyskinesia are considered for subthalamic nucleus (STN) deep brain stimulation (DBS) surgery. Therapeutic DBS leads to a reduction in pathological neuronal synchronization seen in PD. While continuous high-frequency stimulation is effective for ameliorating motor symptoms, the investigators hypothesize that different stimulation patterns which are designed to better target excessive synchrony in a patient-tailored manner, may result in more efficient and effective therapy with fewer side effects. This overarching hypothesis is supported by prior foundational preclinical and clinical research. Medtronic has developed proprietary technology that allows implantable neural stimulators (INS) to deliver both standard clinical electrical stimulation therapy and to record bioelectric data (i.e. local field potentials; LFPs) through DBS leads implanted in the brain. Medtronic's 3rd-generation sensing DBS INS, Percept PC, is FDA-approved for treating PD and can be used to explore unique biomarkers of brain state changes associated with activities of daily living and disease symptomatic states.

This research will use Percept PC INS latent capabilities to deliver research stimulation. Importantly, all stimulation in this research project will be delivered using charge-balanced pulses, in compliance with all FDA safety guidelines including frequency (≤ 250 Hz) and charge density (30 µC/cm2/phase). At the conclusion of the research study, standard clinical stimulation will be re-activated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's Disease who were recommended for STN DBS using standard clinical inclusion and exclusion criteria (e.g., presence of coagulopathy, dementia, untreated depression, pre-existing implanted stimulation system, prior intracranial surgery, history of alcohol or drug abuse)
* Patients have been previously implanted with bilateral STN DBS and the Medtronic Percept PC implantable neural stimulator.
* Patients are optimized for clinical stimulation and medication for at least 3 months post-surgery for the implantation of their DBS system.
* Consent to study participation
* Presence of a robust beta peak (detectable using the Percept BrainSense Survey feature; ≥ 0.7 µV/rtHz), intra-operatively (assessed via Lead Confirm technology from Alpha Omega)
* Good response to stimulation (30% improvement on UPDRS III compared to baseline OFF), at least 3 months post-surgery.

Exclusion Criteria:

* Not currently implanted with the Medtronic Percept INS
* Not willing to participate in the study
* Unstable stimulation with need for frequent reprogramming or further adjustment
* Significant stimulation-induced side effects
* Need for unusual programming parameters such as very high (> 200 Hz) or low (< 100) frequencies (due to cycle limitations)
* The patient has an implanted cardiac device
* The patients Medtronic Percept TM PC indicates elective-replacement-indicated (ERI) at the start of the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of novel DBS stimulation patterns. | Years 1-2
  To assess if the novel stimulation patterns provide similar side effect profile, when compared to standard clinical stimulation, tolerability will be assessed by:
  1. Number of study participants experiencing stimulation-related side effects. Side effects will be measured as patient-reported severity and type of side effect.
  2. Number of study participants experiencing stimulation-related Adverse Events.

SECONDARY OUTCOMES:
Response to novel DBS stimulation patterns. | Years 1-2
  To assess if the novel stimulation patterns provide similar motor symptom benefit, when compared to standard clinical stimulation, response will be assessed by:
  1. UPDRS Part III exam instrumented with inertial sensors will provide severity scores from 0-4 for tremor, bradykinesia, rigidity and dyskinesia.
  2. Balance and gait measures will be obtained by inertial sensors placed in the extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Abosch, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No